CLINICAL TRIAL: NCT06529601
Title: Comparison Between CAD/CAM and Conventional Mandibular Fixed Retainers: a Randomized Controlled Trial
Brief Title: Comparison Between CAD/CAM and Conventional Mandibular Fixed Retainers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LF15
Record Dates: First submitted 2024-07-10; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Orthodontic Retainers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM mandibular fixed retainer (Experimental)
  Interventions: Device: CAD/CAM mandibular fixed retainer
- Conventional mandibular fixed retainer (Active Comparator)
  Interventions: Device: Conventional mandibular fixed retainer

INTERVENTIONS:
Device: CAD/CAM mandibular fixed retainer — Keeppy is a Class IIa custom-made medical device manufactured by Digital Service Leone s.r.l. - via Pratese 160/b, Florence, Italy. The Keeppy is an individualized fixed retainer, made of a Nickel-free Chrome Cobalt alloy, produced with a CAD-CAM procedure starting from a digital impression made with an intraoral optical scanner (3 Shape), which allows a perfect adaptation to the lingual surfaces of the 6 lower anterior teeth on which it is bonded. The device is characterized by the presence of applicators that can be placed temporarily on the buccal surface of the canines, which facilitate the clinician in the precise application of the device and which are removed as soon as the bonding phase of the retainer is complete. Bonding is performed using classic composite resins following a preparation phase of the lingual surface of the tooth consisting of the application of etchant (37% orthophosphoric acid) for 30 seconds and adhesive (primer-bonding).
  Other Names: Keeppy
  Arms: CAD/CAM mandibular fixed retainer
Device: Conventional mandibular fixed retainer — The standard control device, which is among the most commonly used in routine clinical practice, consists of a steel braided wire. The device selected for the Class IIa investigation is the Ortho Flex Tech manufactured by Reliance Orthodontic Products, Inc. 1540 West Thorndale Ave. Itasca, IL 60143 USA. The Ortho Flex Tech steel braided wire is manually shaped by the clinician and cut with a wire cutter so that it has the proper length to extend over the 6 dental elements. Once the correct length has been defined, it is then held in place on the lingual surface of the teeth by the use of 2 interdental wires passing doubly through the interdental area (between the lateral incisor and canine on one side and the other). This allows the device to be bonded using composite resin after etching the lingual surfaces of the lower anterior teeth.
  Arms: Conventional mandibular fixed retainer

SUMMARY:
The devices compared in this study are 'retainers', i.e. fixed orthodontic retainers applied to the lingual surface of the central and lateral incisors and lower canines bilaterally. Their function is to maintain dental alignment once fixed orthodontic therapy has ended. In particular, the CAD/CAM device Keeppy patented by the company Leone SpA (Via Ponte a Quaracchi 50, Sesto Fiorentino, Florence) will be compared with the standard retainer made from a steel braided wire (Ortho FlexTech, Reliance Orthodontic Products Inc., 1540 West Thorndale Ave, Itasca, Illinois, USA).

This is a single-center, national, controlled, superiority, randomized, crossover, open-label study.

The aim of this study is to evaluate whether the CAD/CAM retainer results in fewer failures (fractures or detachments) over a period of 6 months and 2 years compared to the standard retainer. In addition, the aim of the study is to evaluate whether the Keeppy device results in the maintenance of better periodontal health as judged by the use of plaque and bleeding indices on the surfaces of the lower six anterior teeth compared to the standard retainer. Other objectives consist of the patient's assessment of pain, difficulty in speaking and esthetic satisfaction and the stability of the lower anterior tooth sector.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed fixed orthodontic therapy between the ages of 13 and 20 years;
* Patients whose parents will sign the informed consent

Exclusion Criteria:

* Presence of dental anomalies in number (excess or deficiency) in the lower anterior teeth
* Patients with metal allergies.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Retainer failure at 6-month and 2-year follow-ups | At 6 months and at 2 years
  The primary endpoint is retainer failures at 6-month and 2-year follow-ups. Failure is defined as any complication requiring a retainer repair, in particular total or partial detachment and total or partial fracture.

SECONDARY OUTCOMES:
Assessment of the plaque and gingival bleeding index at the central and lateral incisors and lower canines. | At baseline, at 6 months and at 2 years
  Assessment of the plaque and gingival bleeding index at the central and lateral incisors and lower canines.
Pain reported by patients | At baseline, at one month, at 6 months and at 2 years
  Pain measured through Visual Analogue Scale (VAS) with minimum value of 0 and maximum value of 10. Higher scores mean worse pain.
Difficulty in speaking reported by patients | At baseline, at one month, at 6 months and at 2 years
  Difficulty in speaking measured through Visual Analogue Scale (VAS) with minimum value of 0 and maximum value of 10. Higher scores mean worse difficulty in speaking.
Aesthetic satisfaction reported by patients | At baseline, at one month, at 6 months and at 2 years
  Aesthetic satisfaction measured through Visual Analogue Scale (VAS) with minimum value of 0 and maximum value of 10. Higher scores mean higher aesthetic satisfaction.
Stability of the alignment of the lower anterior teeth | At 6 months and at 2 years
  Stability of the alignment of the lower anterior teeth will be assessed with Little's irregularity index and the intercanine diameter measured on the virtual impression of the patient's teeth.